CLINICAL TRIAL: NCT05585138
Title: Effects of Preoperative Segmental Breathing Exercise on Postoperative Pulmonary Complications in Patients Awaiting Coronary Artery Bypass Graft Surgery (CABG)
Brief Title: Effects of Segmental Breathing Exercise in Patients Awaiting Coronary Artery Bypass Graft Surgery (CABG)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/0345 Munaza Tabassum
Record Dates: First submitted 2022-09-15; First posted 2022-10-18 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Complications Due to Coronary Artery Bypass Graft
Keywords: CABG, segmental breathing, pulmonary complications

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Segmental breathing exercise (Experimental): segmental breathing exercise (apical costal expansion exercises, lateral costal expansion exercises, posterior costal expansion exercises) combined with Conventional Treatment ( deep breathing exercise ).
  Group-A (interventional group) will receive segmental breathing exercises for one month 5 days a week and 2 sessions per day for 15 minutes for each patient
  Interventions: Other: segmental breathing exercise; Other: deep breathing
- conventional therapy (Active Comparator): Conventional Treatment (deep breathing exercise). conventional treatment will be for one month 5 days a week 10 to 15 repetitions of deep breathing exercise 2times a day.
  Interventions: Other: deep breathing

INTERVENTIONS:
Other: segmental breathing exercise — Group-A (interventional group) will receive segmental breathing exercises and deep breathing. segmental breathing exercise will be performed by taking a deep and long breath from nose patient inhale air in to lungs and in exhalation therapist will apply pressure on intercostal spaces at apical, lateral and posterior for one month 5 days a week and 2 sessions per day for 15 minutes for each patient. conventional treatment will be for one month 5 days a week 10 to 15 repetitions of deep breathing exercise 2 times a day.
  Arms: Segmental breathing exercise
Other: deep breathing — conventional treatment will be for one month 5 days a week 10 to 15 repetitions of deep breathing exercise 2 times a day. . deep breathing exercise will be performed by taking a deep and long breath from nose patient inhale air in to lungs and will exhale through mouth.

SUMMARY:
To determine the effects of preoperative segmental breathing exercise on postoperative pulmonary complications in patients awaiting coronary artery bypass graft surgery (CABG).

This study will be a randomized controlled trial. This study will be conducted in cardiac surgery department at Faisalabad institute of cardiology. sample size will be 44including both male and female. Non- probability purposive sampling technique will be used.

Modified healthy heart questionnaire will be used as a screening tool. Baseline, postoperatively before discharge at week 5 assessment will be done by 6-minute walk test. Subjects in group A (interventional group) will be treated using segmental breathing exercises combined with Conventional Treatment (deep breathing exercise ) and the group B (control group) will be treated with only conventional treatment. Group-A (interventional group) will receive segmental breathing exercises for one month 5 days a week and 2 sessions per day for 15 minutes for each patient. conventional treatment will be for one month 5 days a week 10 to 15 repetitions of deep breathing exercise 2times a day. Dyspnea will be checked baselineand at week5 by modified Borg scale.Sputum cup was used for expectoration of sputum . Quality of life will be checked baseline and at week 5by SF-12 Questionnaire. Outcome variables will be 6MWT, dyspnea, quality of life, oxygen saturation, heart rate, blood pressure and expectoration of sputum. Data will be analyzed on SPSS-25.

DETAILED DESCRIPTION:
This study will be a randomized controlled trial. This study will be conducted in cardiac surgery department at Faisalabad institute of cardiology. sample size will be 44including both male and female. Non- probability purposive sampling technique will be used.

Modified healthy heart questionnaire will be used as a screening tool. Baseline, postoperatively before discharge at week 5 assessment will be done by 6-minute walk test. Subjects in group A (interventional group) will be treated using segmental breathing exercises combined with Conventional Treatment (deep breathing exercise ) and the group B (control group) will be treated with only conventional treatment. Group-A (interventional group) will receive segmental breathing exercises for one month 5 days a week and 2 sessions per day for 15 minutes for each patient. conventional treatment will be for one month 5 days a week 10 to 15 repetitions of deep breathing exercise 2times a day. Dyspnea will be checked baselineand at week5 by modified Borg scale.Sputum cup was used for expectoration of sputum . Quality of life will be checked baseline and at week 5by SF-12 Questionnaire. Outcome variables will be 6MWT, dyspnea, quality of life, oxygen saturation, heart rate, blood pressure and expectoration of sputum. Data will be analyzed on SPSS-25.

ELIGIBILITY:
Inclusion Criteria:

* patients who will be willing to participate in study
* Patient having age 40 to 65 years of age both male and female
* Diagnosed patients of Double vessel coronary artery disease and Triple vessel coronary artery disease
* Controlled diabetic and hypertensive patients.

Exclusion Criteria:

* patient on bronchodilators.
* Left ventricular ejection fraction< 40 %.
* Valvular disease.
* Patient having dysrhythmias or pacemaker dependent.
* Anemic patient.
* Patient having asthma, chronic obstructive pulmonary disease and interstitial lung disease
* Patient with neurological disorder.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2022-05-02 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-26 (Actual)

PRIMARY OUTCOMES:
Change in 6 minute walk test | baseline and week 5
  The 6 Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.It measures the walking distance of subjects within a fixed time to quantify the functional capacity of the subjects, which refers to the total distance the subjects walked within 6 minutes.
Change in Modified Borg Dyspnea Scale | baseline and week 5
  The Modified Borg Dyspnea Scale (MBS) is a 0 to 10 rated numerical score used to measure dyspnea as reported by the patient during submaximal exercise and is routinely administered during six-minute walk testing (6MWT). It starts at number 0 where your breathing is causing you no difficulty at all and progresses through to number 10 where your breathing difficulty is maximal.
Change in short form-12 Health related quality of life questionnaire | baseline and week 5
  It is a self-reported outcome measure assessing the impact of health on an individual's everyday life. The SF-12v2 is a health-related quality-of-life questionnaire consisting of twelve questions that measure eight health domains to assess physical and mental health. Physical health-related domains include General Health (GH), Physical Functioning (PF), Role Physical (RP), and Body Pain (BP). short form-12 questionnaire will be used to measure quality of life in CABG patients. Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Sumera Abdul Hameed, MS, Principal Investigator — Riphah International University
Locations (1):
- Faisalabad institute of cardiology, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Caliskan E, de Souza DR, Boning A, Liakopoulos OJ, Choi YH, Pepper J, Gibson CM, Perrault LP, Wolf RK, Kim KB, Emmert MY. Saphenous vein grafts in contemporary coronary artery bypass graft surgery. Nat Rev Cardiol. 2020 Mar;17(3):155-169. doi: 10.1038/s41569-019-0249-3. Epub 2019 Aug 27. PMID 31455868
- [Background] Yang J, Biery DW, Singh A, Divakaran S, DeFilippis EM, Wu WY, Klein J, Hainer J, Ramsis M, Natarajan P, Januzzi JL, Nasir K, Bhatt DL, Di Carli MF, Blankstein R. Risk Factors and Outcomes of Very Young Adults Who Experience Myocardial Infarction: The Partners YOUNG-MI Registry. Am J Med. 2020 May;133(5):605-612.e1. doi: 10.1016/j.amjmed.2019.10.020. Epub 2019 Nov 9. PMID 31715169
- [Background] Pooria A, Pourya A, Gheini A. Postoperative complications associated with coronary artery bypass graft surgery and their therapeutic interventions. Future Cardiol. 2020 Sep;16(5):481-496. doi: 10.2217/fca-2019-0049. Epub 2020 Jun 4. PMID 32495650
- [Background] Thybo Karanfil EO, Moller AM. Preoperative inspiratory muscle training prevents pulmonary complications after cardiac surgery - a systematic review. Dan Med J. 2018 Mar;65(3):A5450. PMID 29510803
- [Background] Chen JO, Liu JF, Liu YQ, Chen YM, Tu ML, Yu HR, Lin MC, Lin CC, Liu SF. Effectiveness of a perioperative pulmonary rehabilitation program following coronary artery bypass graft surgery in patients with and without COPD. Int J Chron Obstruct Pulmon Dis. 2018 May 16;13:1591-1597. doi: 10.2147/COPD.S157967. eCollection 2018. PMID 29805258
- [Background] Gomes Neto M, Martinez BP, Reis HF, Carvalho VO. Pre- and postoperative inspiratory muscle training in patients undergoing cardiac surgery: systematic review and meta-analysis. Clin Rehabil. 2017 Apr;31(4):454-464. doi: 10.1177/0269215516648754. Epub 2016 Jul 10. PMID 27154820
- [Background] Cordeiro AL, de Melo TA, Neves D, Luna J, Esquivel MS, Guimaraes AR, Borges DL, Petto J. Inspiratory Muscle Training and Functional Capacity in Patients Undergoing Cardiac Surgery. Braz J Cardiovasc Surg. 2016 Apr;31(2):140-4. doi: 10.5935/1678-9741.20160035. PMID 27556313
- [Background] Alaparthi GK, Amin R, Gatty A, Raghavan H, Bairapareddy KC, Vaishali K, Borghi-Silva A, Hegazy FA. Contrasting effects of three breathing techniques on pulmonary function, functional capacity and daily life functional tasks in patients following valve replacement surgery- A pilot randomized clinical trial. Heliyon. 2021 Jul 22;7(7):e07643. doi: 10.1016/j.heliyon.2021.e07643. eCollection 2021 Jul. PMID 34377862
- [Background] Sahar W, Ajaz N, Haider Z, Jalal A. Effectiveness of Pre-operative Respiratory Muscle Training versus Conventional Treatment for Improving Post operative Pulmonary Health after Coronary Artery Bypass Grafting. Pak J Med Sci. 2020 Sep-Oct;36(6):1216-1219. doi: 10.12669/pjms.36.6.2899. PMID 32968383
- [Background] Moradian ST, Heydari AA, Mahmoudi H. What is the Role of Preoperative Breathing Exercises in Reducing Postoperative Atelectasis after CABG? Rev Recent Clin Trials. 2019;14(4):275-279. doi: 10.2174/1574887114666190710165951. PMID 31291879
- [Background] Zolfaghari M, Mirhosseini SJ, Baghbeheshti M, Afshani A, Moazzam S, Golabchi A. Effect of physiotherapy on quality of life after coronary artery bypass graft surgery: A randomized study. J Res Med Sci. 2018 Jun 6;23:56. doi: 10.4103/jrms.JRMS_96_17. eCollection 2018. PMID 30057640
- [Background] Pehlivan E, Turna A, Gurses A, Gurses HN. The effects of preoperative short-term intense physical therapy in lung cancer patients: a randomized controlled trial. Ann Thorac Cardiovasc Surg. 2011;17(5):461-8. doi: 10.5761/atcs.oa.11.01663. Epub 2011 Jul 13. PMID 21881371
- [Background] Matheus GB, Dragosavac D, Trevisan P, Costa CE, Lopes MM, Ribeiro GC. Inspiratory muscle training improves tidal volume and vital capacity after CABG surgery. Rev Bras Cir Cardiovasc. 2012 Jul-Sep;27(3):362-9. doi: 10.5935/1678-9741.20120063. English, Portuguese. PMID 23288176
- [Background] Savci S, Degirmenci B, Saglam M, Arikan H, Inal-Ince D, Turan HN, Demircin M. Short-term effects of inspiratory muscle training in coronary artery bypass graft surgery: a randomized controlled trial. Scand Cardiovasc J. 2011 Oct;45(5):286-93. doi: 10.3109/14017431.2011.595820. Epub 2011 Jul 27. PMID 21793631
- [Background] Chen YC, Chen KC, Lu LH, Wu YL, Lai TJ, Wang CH. Validating the 6-minute walk test as an indicator of recovery in patients undergoing cardiac surgery: A prospective cohort study. Medicine (Baltimore). 2018 Oct;97(42):e12925. doi: 10.1097/MD.0000000000012925. PMID 30335028
- [Background] Failde I, Medina P, Ramirez C, Arana R. Construct and criterion validity of the SF-12 health questionnaire in patients with acute myocardial infarction and unstable angina. J Eval Clin Pract. 2010 Jun;16(3):569-73. doi: 10.1111/j.1365-2753.2009.01161.x. Epub 2010 Apr 21. PMID 20438603
- [Background] Pacaric S, Turk T, Eric I, Orkic Z, Petek Eric A, Milostic-Srb A, Farcic N, Barac I, Nemcic A. Assessment of the Quality of Life in Patients before and after Coronary Artery Bypass Grafting (CABG): A Prospective Study. Int J Environ Res Public Health. 2020 Feb 22;17(4):1417. doi: 10.3390/ijerph17041417. PMID 32098322
- [Background] Reychler G, Beaumont M, Latiers AC, Pieters T, Fremault A. Dyspnea could be accurately assessed by a caregiver in hospitalized patients with respiratory diseases: Interrater reliability and agreement study. Braz J Phys Ther. 2021 Nov-Dec;25(6):735-740. doi: 10.1016/j.bjpt.2021.04.010. Epub 2021 May 24. PMID 34119444